CLINICAL TRIAL: NCT01118650
Title: Concordance of the Quotient ADHD System Report With Teacher and Parent Assessments in School-Aged Children Receiving an Individualized Education Program (IEP) or 504 Accommodations in the Classroom Setting for Symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Concordance of the Quotient Attention Deficit Hyperactivity Disorder (ADHD) System Report With Teacher and Parent Assessments for Symptoms of ADHD
Status: Withdrawn | Type: Observational
Why Stopped: No interest from school district
Sponsor: BioBehavioral Diagnostics Company (Industry)
Collaborators: New Hampshire School Administrative Unit #44 (Unknown)
Responsible Party: Sponsor
Other Study IDs: BBD0108
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Inattention; Hyperactivity; Impulsivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Impulsive Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To demonstrate concordance between the Quotient ADHD System Report and standard DSM-IV based parent and teacher reported rating/assessment scales, currently the accepted method of symptom measurement for subjects diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
Public school based study for children ages 8 through 14 years of age.

Children previously identified and currently receiving an Individualized Education Program (IEP) or 504 accommodations in the classroom setting for symptoms of ADHD.

Open enrollment of 30 subjects, both male and female.

One study visit in which subjects will perform/receive the following assessments/evaluations:

1. Quotient ADHD System Test
2. Vanderbilt ADHD Diagnostic Teacher Rating Scale
3. Vanderbilt ADHD Diagnostic Parent Rating Scale

The primary analytical goal is to examine the extent of agreement of the Quotient ADHD System(either individual measures or in combination) with standard measures (Vanderbilt ADHD Diagnostic Teacher Rating Scale and Vanderbilt ADHD Diagnostic Parent Rating Scale) and to compare this agreement with that seen between the standard measures.

ELIGIBILITY:
Inclusion Criteria:

* A student attending one of three public elementary schools in the New Hampshire School Administrative Unit #44.
* Age 8 through 14 years old at time of enrollment.
* Pre-identified as receiving an Individualized Education Program (IEP) or 504 accommodations for symptoms of ADHD in the school setting by the Special Education Coordinator in the school district.
* A parent/guardian of the child must be willing to participate.

Exclusion Criteria:

* No subject will be excluded from participation based on race, ethnicity, or gender. Anyone meeting inclusion criteria, who are willing to sign consent and participate, will be included in the study.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Public School based study for children ages 8 through 14 years of age who have been identified and are currently receiving an Individualized Education Program (IEP) or 504 accommodations in the classroom setting for symptoms of Attention Deficit Hyperactivity Disorder
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calvin R Sumner, MD, Principal Investigator — BioBehavioral Diagnostic Company